CLINICAL TRIAL: NCT00089674
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate AMG 162 in the Treatment of Bone Loss in Subjects Undergoing Androgen-Deprivation Therapy for Non-metastatic Prostate Cancer
Brief Title: AMG 162 in the Treatment of Bone Loss in Subjects Undergoing Androgen-Deprivation Therapy for Non-metastatic Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20040138; HALT Prostate Cancer
Record Dates: First submitted 2004-08-09; First posted 2004-08-11 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Bone Loss with Prostate Cancer; Treatment of bone loss in patients undergoing androgen deprivation therapy (ADT) for non-metastatic prostate cancer (PC).
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AMG 162 (Experimental)
  Interventions: Drug: AMG 162
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 162 — 60 mg (1.0mL) administered subcutaneously at Day 1, Months 6, 12, 18, 24, 30
  Arms: AMG 162
Drug: Placebo — 60 mg (1.0mL) administered subcutaneously at Day 1, Months 6, 12, 18, 24, 30
  Arms: Placebo

SUMMARY:
This study will evaluate AMG 162 in the treatment of bone loss in subjects undergoing Androgen-Deprivation Therapy for Non-metastatic Prostate Cancer.

ELIGIBILITY:
Other criteria also apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1468 (Actual)
Dates: Start 2004-08-01 (Actual); Primary Completion 2008-05-16 (Actual); Study Completion 2010-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Egerdie RB, Saad F, Smith MR, Tammela TL, Heracek J, Sieber P, Ke C, Leder B, Dansey R, Goessl C. Responder analysis of the effects of denosumab on bone mineral density in men receiving androgen deprivation therapy for prostate cancer. Prostate Cancer Prostatic Dis. 2012 Sep;15(3):308-12. doi: 10.1038/pcan.2012.18. PMID 22641239
- [Background] Lippuner k, Wolff JM, Hadji P, Braun A, Ke C, Steinle T, Eisen C. Risk reduction for vertebral fractures in patients with normal to osteopenic bone mineral density receiving denosumab: A subgroup analysis of the HALT Prostate Cancer Trial. Osteologie 2014;23(2):117-122. [published in German only]
- [Background] Smith MR, Egerdie B, Hernandez Toriz N, Feldman R, Tammela TL, Saad F, Heracek J, Szwedowski M, Ke C, Kupic A, Leder BZ, Goessl C; Denosumab HALT Prostate Cancer Study Group. Denosumab in men receiving androgen-deprivation therapy for prostate cancer. N Engl J Med. 2009 Aug 20;361(8):745-55. doi: 10.1056/NEJMoa0809003. Epub 2009 Aug 11. PMID 19671656
- [Background] Smith MR, Saad F, Egerdie B, Sieber P, Tammela TLj, Leder BZ, Ke C, Goessl C. Denosumab and changes in bone turnover markers during androgen deprivation therapy for prostate cancer. J Bone Miner Res. 2011 Dec;26(12):2827-33. doi: 10.1002/jbmr.492. PMID 21898590
- [Background] Smith MR, Saad F, Egerdie B, Szwedowski M, Tammela TL, Ke C, Leder BZ, Goessl C. Effects of denosumab on bone mineral density in men receiving androgen deprivation therapy for prostate cancer. J Urol. 2009 Dec;182(6):2670-5. doi: 10.1016/j.juro.2009.08.048. PMID 19836774
- [Derived] Kuchler U, Luvizuto ER, Tangl S, Watzek G, Gruber R. Short-term teriparatide delivery and osseointegration: a clinical feasibility study. J Dent Res. 2011 Aug;90(8):1001-6. doi: 10.1177/0022034511407920. Epub 2011 May 9. PMID 21555773
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Enrolled: 15-Apr-2004 Last Subject Enrolled: 29-Apr-2005
Groups:
- Placebo: Placebo administered subcutaneous every 6 months for 3 years
- Denosumab 60 mg Q6M: Denosumab 60 mg administered subcutaneous (SC) every 6 months for 3 years
Period: Overall Study
Arm/Group | Placebo | Denosumab 60 mg Q6M
Started | 734 | 734
Received Study Drug | 730 | 726
Completed | 445 | 467
Not Completed | 289 | 267
Not completed — Physician Decision | 4 | 2
Not completed — Adverse Event | 23 | 29
Not completed — Withdrawal by Subject | 143 | 127
Not completed — Death | 43 | 43
Not completed — Disease progression | 21 | 23
Not completed — Ineligibility determined | 8 | 10
Not completed — Lost to Follow-up | 21 | 17
Not completed — Noncompliance | 7 | 3
Not completed — Other | 5 | 9
Not completed — Requirement for alternative therapy | 14 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Denosumab 60 mg Q6M | Total
Number analyzed (Participants) | 734 | 734 | 1468
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.5 (7.1) | 75.3 (7) | 75.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 734 | 734 | 1468
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 3 | 5 | 8
  Japanese | 4 | 1 | 5
  American Indian or Alaska Native | 2 | 0 | 2
  Other | 3 | 0 | 3
  White or Caucasian | 609 | 615 | 1224
  Black or African American | 32 | 36 | 68
  Hispanic or Latino | 81 | 77 | 158

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 24
Description: Lumbar Spine Bone Mineral Density Percent Chnage From Baseline at Month 24 Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 24 months
Population: Randomized subjects who had a nonmissing baseline and >= 1 nonmissing postbaseline data before or at month 24. LOCF used as imputation method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 716 | 714
Percent Change from Baseline | -1 [-1.4 to -0.7] | 5.6 [5.3 to 5.9]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 6.7, 95% CI [6.2 to 7.1]

2. Secondary Outcome: Femoral Neck Bone Mineral Density Percent Change From Baseline at Month 24
Description: Femoral Neck Bone Mineral Density Percent Change From Baseline at Month 24 Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 24 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 706 | 701
Percent Change from Baseline | -1.5 [-1.8 to -1.1] | 2.4 [2.1 to 2.8]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA — Adjusted for multiplicity using the prespecified hierarchical analysis strategy and Hochberg procedure; Mean Difference (Final Values) = 3.9, 95% CI [3.5 to 4.4]

3. Secondary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 24
Description: Total Hip Bone Mineral Density Percent Change From Baseline at Month 24 Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 24 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 706 | 701
Percent Change from Baseline | -2 [-2.3 to -1.8] | 2.7 [2.5 to 3.0]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA — Adjusted for multiplicity using the prespecified hierarchical analysis strategy and Hochberg procedure; Mean Difference (Final Values) = 4.8, 95% CI [4.4 to 5.1]

4. Secondary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 36
Description: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 36 Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 36 months
Population: Randomized subjects who had a nonmissing baseline and >= 1 nonmissing postbaseline data before or at month 36. LOCF used as imputation method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 716 | 714
Percent Change from Baseline | -1.2 [-1.5 to -0.8] | 6.8 [6.4 to 7.1]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA — Adjusted for multiplicity using the prespecified hierarchical analysis strategy and Hochberg procedure; Mean Difference (Final Values) = 7.9, 95% CI [7.4 to 8.4]

5. Secondary Outcome: Femoral Neck Bone Mineral Density Percent Change From Baseline at Month 36
Description: Femoral Neck Bone Mineral Density Percent Change From Baseline at Month 36 Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 36 months
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 706 | 701
Percent Change from Baseline | -1.8 [-2.2 to -1.5] | 3 [2.7 to 3.4]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA — Adjusted for multiplicity using the prespecified hierarchical analysis strategy and Hochberg procedure; Mean Difference (Final Values) = 4.9, 95% CI [4.4 to 5.4]

6. Secondary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 36
Description: Total Hip Bone Mineral Density Percent Change From Baseline at Month 36 Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 36 months
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 706 | 701
Percent Change from Baseline | -2.6 [-2.8 to -2.3] | 3.2 [2.9 to 3.4]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA — Adjusted for multiplicity using the prespecified hierarchical analysis strategy and Hochberg procedure; Mean Difference (Final Values) = 5.7, 95% CI [5.4 to 6.1]

7. Secondary Outcome: Number of Participants With Any Fracture Through Month 36
Description: Any fracture includes osteroporotic fractures at any site excluding skull, facial, mandible, metacarpals, finger phalanges, and toe phalanges.
Time Frame: 36 months
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 734 | 734
Participants | 53 | 38
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.1048, Regression, Logistic — Adjusted for multiplicity using the prespecified hierarchical analysis strategy and Hochberg procedure; Odds Ratio (OR) = 0.7, 95% CI [0.46 to 1.08]

8. Secondary Outcome: Number of Participants With a New Vertebral Fracture Through Month 36
Description: New Vertebral Fracture Assessed by Lateral Spine X-ray using Genant Semiquantitative Scoring Method excluding any symptomatic new vertebral fracture associated with high trauma severity or a pathologic fracture.
Time Frame: 36 months
Population: All randomized subjects who have a baseline and >= 1 postbaseline evaluation of vertebral fracture at or before 3 years.
Measure: Number; unit: Participants
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 673 | 679
Participants | 26 | 10
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.0125, Regression, Logistic — Adjusted for multiplicity using the prespecified hierarchical analysis strategy and Hochberg procedure; Odds Ratio (OR) = 0.37, 95% CI [0.18 to 0.78]

9. Secondary Outcome: Time to First Clinical Fracture Through Month 36
Description: A clinical fracture was defined as any nonvertebral fracture or clinically evident fracture at the cervical vertebrae, thoracic vertebrae, and lumbar vertebrae that was associated with signs and/or symptoms indicative of a fracture. Fractures associated with high trauma severity and pathologic (ie, metastatic) fractures were excluded. Since the median time was not reached, time to first clinical fracture is represented by the Kaplan-Meier estimate of the percentage of participants with a clinical fracture.
Time Frame: 36 months
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 734 | 734
Percentage of participants | 5.2 | 4.7
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.7961, Regression, Cox — Adjusted for multiplicity using the prespecified hierarchical analysis strategy and Hochberg procedure; Hazard Ratio (HR) = 0.94, 95% CI [0.57 to 1.55]

10. Secondary Outcome: Number of Participants With Any Fracture Through Month 24
Description: as for outcome 7
Time Frame: 24 months
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 734 | 734
Participants | 45 | 32
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.7961, Regression, Logistic — Adjusted for multiplicity using the prespecified hierarchical analysis strategy and Hochberg procedure; Odds Ratio (OR) = 0.7, 95% CI [0.44 to 1.11]

ADVERSE EVENTS:
Time Frame: 36 months
Description: Five participants randomized to placebo received 1 dose of denosumab in error and are included in the denosumab group for safety analysis. The table of Other Adverse Events summarizes non-serious occurrences of adverse events that exceeded a 5% frequency in either treatment arm.
Arm/Group | Placebo | Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 222/725 | 253/731
Other Adverse Events (participants affected / at risk) | 364/725 | 390/731
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=725) | Denosumab 60 mg Q6M (N=731)
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 3 | 4
Acute myocardial infarction (Cardiac disorders) | 5 | 4
Angina pectoris (Cardiac disorders) | 4 | 4
Angina unstable (Cardiac disorders) | 3 | 1
Aortic valve disease (Cardiac disorders) | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 8 | 11
Atrial flutter (Cardiac disorders) | 2 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 3 | 4
Cardiac arrest (Cardiac disorders) | 4 | 4
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 4
Cardiac failure congestive (Cardiac disorders) | 10 | 6
Cardiac flutter (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 2
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 11 | 9
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial fibrosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 18 | 14
Myocardial ischaemia (Cardiac disorders) | 6 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 5
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Trifascicular block (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 2
Glaucoma (Eye disorders) | 1 | 1
Retinal detachment (Eye disorders) | 0 | 2
Retinal vascular thrombosis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 2 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 3 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 2 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 2
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Leukoplakia oral (Gastrointestinal disorders) | 0 | 1
Lumbar hernia (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Peritoneal disorder (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 3 | 2
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 4 | 0
Condition aggravated (General disorders) | 1 | 0
Death (General disorders) | 5 | 2
Gait disturbance (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 5
Oedema peripheral (General disorders) | 2 | 1
Pelvic mass (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Sudden death (General disorders) | 1 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 4
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 4
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 2
Bronchopneumonia (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Bursitis infective staphylococcal (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 4 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 5
Endocarditis bacterial (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal gangrene (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 3
Localised infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 11 | 11
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1
Prostate infection (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 2
Pseudomonas infection (Infections and infestations) | 0 | 1
Pyothorax (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 0
Septic shock (Infections and infestations) | 4 | 0
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Urosepsis (Infections and infestations) | 2 | 3
Viral infection (Infections and infestations) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Device failure (Injury, poisoning and procedural complications) | 1 | 0
Failure of implant (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 2
Femur fracture (Injury, poisoning and procedural complications) | 2 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 2
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 2
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Nerve root injury cervical (Injury, poisoning and procedural complications) | 0 | 1
Pacemaker complication (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 5
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 3
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Stenosis of vesicourethral anastomosis (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 3 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 6
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 3
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Brain injury (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 3
Cerebral infarction (Nervous system disorders) | 2 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 12 | 10
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Cerebrovascular spasm (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 3
Hemiparesis (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1
Hypoxic encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1
Senile dementia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 8
Syncope vasovagal (Nervous system disorders) | 1 | 1
Thalamus haemorrhage (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 4 | 9
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 3
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 2
Hallucination (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 1 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 1 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Contracted bladder (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Polyuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 4
Renal failure acute (Renal and urinary disorders) | 5 | 3
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 2
Ureteric perforation (Renal and urinary disorders) | 0 | 1
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 6
Urinary tract disorder (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1
Hernia repair (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Implantable defibrillator replacement (Surgical and medical procedures) | 0 | 1
Kidney ablation (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Spinal operation (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 3 | 2
Aortic dissection (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Cardiovascular insufficiency (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 4
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 5 | 4
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 5
Hypovolaemic shock (Vascular disorders) | 0 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 3
Peripheral artery aneurysm (Vascular disorders) | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 2
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 2
Venous occlusion (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=725) | Denosumab 60 mg Q6M (N=731)
Constipation (Gastrointestinal disorders) | 74 | 73
Diarrhoea (Gastrointestinal disorders) | 39 | 39
Fatigue (General disorders) | 45 | 44
Oedema peripheral (General disorders) | 47 | 52
Nasopharyngitis (Infections and infestations) | 45 | 47
Urinary tract infection (Infections and infestations) | 30 | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 79 | 91
Back pain (Musculoskeletal and connective tissue disorders) | 73 | 79
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 26 | 40
Pain in extremity (Musculoskeletal and connective tissue disorders) | 51 | 66
Dizziness (Nervous system disorders) | 31 | 41
Hot flush (Vascular disorders) | 32 | 38
Hypertension (Vascular disorders) | 47 | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.